CLINICAL TRIAL: NCT02278991
Title: A Prospective, Multicenter, Single-Arm, Post-Market Study Using the Lutonix Drug Coated Balloon for Post-Dilatation of the Bard LifeStent Vascular Stent for Treatment of Long Lesions in Femoropopliteal Arteries
Brief Title: Bard LifeStent and Lutonix DCB for Treatment of Long Lesions in Femoropopliteal Arteries
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: CL0022-01
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lutonix Drug Coated Balloon: Paclitaxel coated balloon catheter
  Interventions: Device: Lutonix Drug Coated Balloon

INTERVENTIONS:
Device: Lutonix Drug Coated Balloon — Subject will receive treatment with the Lutonix Drug Coated Balloon

SUMMARY:
Objective of this study is to evaluate the safety and efficacy of Lutonix 035 Drug Coated Dilatation PTA Catheter with Bard LifeStent Vascular Stent (hereinafter referred to as LifeStent) for treatment of long (10-24 cm) lesions in the SFA and/or proximal popliteal artery.

DETAILED DESCRIPTION:
The study will observe subjects presenting with claudication or ischemic rest pain (Rutherford category 2-4) and long (10-24 cm in length) native lesions in the infra-inguinal segment (superficial femoral artery [SFA] and/or proximal popliteal artery) who are candidates for stenting and pre-/post-dilatation with Drug Coated Balloon (DCB).

ELIGIBILITY:
Inclusion Criteria: Subjects will be included if all of the following inclusion criteria apply:

1. Age ≥18 years;
2. The subject is legally competent and able to understand the information on the study, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, and has duly signed the Informed Consent Form (ICF);
3. Rutherford Category 2-4;
4. Target de novo lesion(s) or non-stented restenotic lesion(s) has angiographic evidence of ≥50% stenosis or occlusion (by visual estimate) and is amenable to treatment with LifeStent® and Lutonix DCB;
5. Patients must be able to be treated with Lutonix DCB and LifeStent®;
6. Total Lutonix DCB treated segment(s) of 10-24 cm in length;
7. Target vessel reference diameter is 4.0-7.0 mm (by visual estimate) and able to be treated with available device size matrix;
8. At least one patent native outflow artery to the ankle free from significant lesion (≥50% stenosis) as confirmed by angiography (treatment of outflow disease is NOT permitted; treatment of in-flow disease is permitted prior to treatment with LifeStent®).
9. No other prior vascular interventions (including contralateral limb) within 2 weeks before and/or planned 30 days after the protocol treatment, with the exception of remote common femoral patch angioplasty separated by at least 2 cm from the target lesion;
10. Female subjects of childbearing potential have a negative urine or serum pregnancy test within 7 days prior to index procedure;
11. Lesion location starts ≥1 cm below the common femoral bifurcation and terminates distally ≤2 cm below the tibial plateau AND ≥1 cm above the origin of the tibioperoneal trunk.

Exclusion Criteria:

1. Pregnant, lactating, or planning on becoming pregnant or men intending to father children;
2. Contraindication to Lutonix DCB or LifeStent® per current IFU;
3. Life expectancy of <1 year;
4. Inability to take required antiplatelet/anticoagulant medications per the LifeStent® and Lutonix DCB IFU, or known contraindication (including allergic reaction) or sensitivity to contrast media, nickel, titanium or tantalum that cannot be adequately managed with pre- and post-procedure medication;
5. Intended treatment of outflow disease during the index procedure;
6. Intended use of laser, atherectomy or cryoplasty during index procedure;
7. Sudden symptom onset, acute vessel occlusion, or acute or subacute thrombus in target vessel;
8. History of stroke within 3 months;
9. History of myocardial infarction, thrombolysis or angina within 2 weeks of enrollment;
10. Participation in an investigational drug or another investigational device study until this study's (Lutonix LifeStent® Study) primary endpoint is reached or previous enrollment in this study;
11. Another medical condition, which, in the opinion of the Investigator, may cause the patient to be noncompliant with the CIP or confound data interpretation;
12. Target vessel and/or lesion involves a previously placed stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital Patients
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Primary patency at 12 months. | 12 months
  Primary patency is defined as the absence of target lesion restenosis and freedom from target lesion revascularization.
Freedom from the composite endpoint of death, index limb amputation, and target vessel revascularization at 30 days. | 30 days
  Freedom from the composite endpoint of death, index limb amputation, and target vessel revascularization at 30 days.

SECONDARY OUTCOMES:
Procedural success | Immediately after Intervention
  Defined as attainment of ≤30% residual stenosis by quantitative angiography immediately after intervention in the absence of peri-procedural complications.
Technical success | Immediately after intervention
  Defined as attainment of ≤30% residual stenosis by quantitative angiography.
Device success | Immediately after intervention
  Defined as successful delivery of the DCB to the target lesion and performance when used according to the clinical investigational plan.
Freedom from Target Lesion Revascularization after 30 days, and 6, 12 and 24 months post-index procedure. | 30 days, 6, 12 and 24 months
  Absence of Target Lesion Revascularization.
Freedom from TVR after 30 days, and 6, 12 and 24 months post-index procedure. | 30 days, 6, 12 and 24 months
  Absence of Target Vessel Revascularization.
Change in resting ankle brachial index (ABI) from baseline to 30 days, and 6, 12 and 24 months post-index procedure | 30 days, 6, 12 and 24 months
  The ABI values will be recorded and compared to the baseline values. The ABI is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm. A ratio of 0.9-1.3 is in the normal range. Lower ratios indicate bad blood perfusion of the leg.
Change in Rutherford Classification from baseline to 30 days, and 6, 12 and 24 months post-index procedure | 30 days, 6, 12 and 24 months
  Patients are enrolled with a Rutherford grade of 2-4 for their target leg. The Rutherford scale is an indicator for the severity of Peripheral Vascular Disease: 0 = no symptoms, 6 = functional foot is no longer salvageable (leading to foot amputation).
All-cause death | 30 days, 6, 12 and 24 months
  Death by any cause will be counted.
Amputation (above the ankle)-free survival | 30 days, 6, 12 and 24 months
  Amputations above the ankle of the target leg will be counted.
Target limb reintervention for treatment of thrombosis of target vessel or embolization to its distal vasculature | 30 days, 6, 12 and 24 months
  Thrombosis in the target vessel and embolizations below the target lesion will be analazed separately from other stenoses.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, Prof., Principal Investigator
Locations (12):
- Germany (10):
  - Klinikum Arnsberg, Arnsberg
  - Herz- und Gefäßzentrum Bad Bevensen, Bad Bevensen
  - Universitäts-Herzzentrum Freiburg Bad Krozingen, Bad Krozingen
  - Angiologikum Hamburg, Hamburg
  - Klinik Immenstadt, Immenstadt im Allgäu
  - Klinikum Kassel, Kassel
  - UKSH - Campus Lübeck, Lübeck
  - RoMed Klinikum Rosenheim, Rosenheim
  - Gefäßzentrum Sonneberg, Sonneberg
  - Klinikum Weiden, Weiden
- University General Hospital of Patras, Pátrai, Greece
- SPZOZ Sanok, Sanok, Poland

IPD SHARING:
Plan to Share IPD: No